CLINICAL TRIAL: NCT05187117
Title: CAPABLE Family Pilot
Brief Title: CAPABLE Family Pilot - Adapting CAPABLE for Older Adults With Mild Cognitive Impairment (MCI)/Early Stage Dementia and Their Care Partners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency); The Rita and Alex Hillman Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00290674
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Dementia, Mild; Mild Cognitive Impairment; Disability Physical; Impairment, Cognitive; Caregiver Burden; Quality of Life; Depression
Keywords: Activities of Daily Living; Instrumental Activities of Daily Living; Caregiving; Physical Function; Executive Function; Home; Intervention; Mild Cognitive Impairment; Early Dementia
MeSH Terms: conditions — Dementia; Lymphoma, Follicular; Cognitive Dysfunction; Caregiver Burden; Depression

STUDY DESIGN:
Intervention Model Description: Waitlist Control Trial
Who Masked: Outcomes Assessor
Masking Description: The assessment collector will be blinded as to whether a participant is in the intervention or waitlist group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Open Label Pilot (Experimental): The Open Label Pilot (Phase 4) will include testing the CAPABLE Family intervention with 6 individuals with MCI or early-stage dementia. At least 5 of the 6 older adults will be required to have a family member involved. Assuming all have a family member involved (though one may not), 12 participants will be enrolled in the open label pilot.
  Open label pilot participants will be asked to provide feedback halfway through the intervention and at the end via phone conversations with the research study team, allowing the study team to make changes accordingly.
  Interventions: Behavioral: CAPABLE Family - Open Label Pilot
- Randomized Control Pilot - Intervention Arm (Experimental): After the open label pilot, 17 older adults (and if available, care partners) will be randomized to the CAPABLE Family intervention. They will be assessed at baseline, after the 4 month intervention, and after the waitlist control arm.
  Interventions: Behavioral: CAPABLE Family - Randomized Control Trial
- Randomized Control Pilot - Waitlist Control Arm (Active Comparator): The waitlist control group, 17 older adults and if available, care partners, will receive the intervention after they have served as controls to the immediate treatment group, ensuring all participants have access to the intervention.
  Interventions: Behavioral: CAPABLE Family - Randomized Control Trial

INTERVENTIONS:
Behavioral: CAPABLE Family - Open Label Pilot — As in CAPABLE (NA_00031539), the delivery characteristics of CAPABLE Family consist of an assessment-driven, individually tailored package of interventions delivered over the course of 4 months by an occupational therapist (OT) (~6 home visits for ≤ 1hour), a registered nurse (RN) (~4 home visits for ≤ 1hour) and a handy worker (HW).
  Adaptations for cognitive decline will be made on a per-client basis as part of the open-label pilot. Topics of adaptations include problem areas addresses, care partner involvement, length/frequency of visits, types of assessments and questions asked, and brainstorming/action planning structure.
  Arms: Open Label Pilot
Behavioral: CAPABLE Family - Randomized Control Trial — As in CAPABLE (NA_00031539), the delivery characteristics of CAPABLE Family consist of an assessment-driven, individually tailored package of interventions delivered over the course of 4 months by an occupational therapist (OT) (~6 home visits for ≤ 1hour), a registered nurse (RN) (~4 home visits for ≤ 1hour) and a handy worker (HW). Refinements based on the open label pilot results will be included.
  Arms: Randomized Control Pilot - Intervention Arm; Randomized Control Pilot - Waitlist Control Arm

SUMMARY:
The purpose of this study is to test the adapted protocol, CAPABLE Family which builds upon the evidenced based CAPABLE program to address older adults with co-occurring physical disability and mild cognitive impairment or early stage dementia and the older adults' caregivers. It will consist of two phases - an open label pilot and waitlist control trial.

DETAILED DESCRIPTION:
CAPABLE (NA_00031539) is an evidence-based program that reduces physical disability, but was designed for people who are cognitively intact.

The investigators seek to adapt CAPABLE to meet the needs of older adults with physical disability and mild cognitive impairment and early stage dementia. The investigators also seek to meet the needs of family members who serve as informal caregivers in relation to the physical function of those with cognitive impairment. The purpose of this pilot study is to test a new protocol for a new program, CAPABLE Family, to address older adults with co-occurring physical disability and dementia and the older adults' caregivers.

CAPABLE is a multicomponent goal-directed program that reduces physical disability by working with the person and environment, but was designed for people who are cognitively intact. Based on the Centers for Medicare and Medicaid (CMS) request, the investigators' team briefly included people with mild dementia in the regular CAPABLE protocol. Looking back on that preliminary data, the investigators identified a subset of 12 older adults with mild dementia with Mini-Mental State Examination (MMSE) scores of 23 or below. The investigators found that more than half improved in Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL) which is promising but much lower than CAPABLE the rest of the cohorts which suggests the need to adapt CAPABLE for people with dementia. Therefore, the investigators have adapted CAPABLE for people with mild cognitive impairment or early stage dementia calling it CAPABLE Family.

As in CAPABLE (NA_00031539), the delivery characteristics of CAPABLE Family consist of an assessment-driven, individually tailored package of interventions delivered over the course of 4 months by an occupational therapist (OT) (~6 home visits for ≤ 1hour), a registered nurse (RN) (~4 home visits for ≤ 1hour) and a handy worker (HW).

This research study is a continuation of IRB00243117 during which the investigators conducted preliminary activities to design the CAPABLE Family intervention. This study will include two phases, an open label pilot and a randomized control trial. The investigators will collect feedback during the open label pilot from the study team clinicians, older adult participants and care partners to further refine the intervention that will be tested as part of the randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* Have at least 1 ADL disability
* Have mild cognitive impairment or mild dementia (as indicated by clinician diagnosis, subjective cognitive complaints, or Blind/Telephone Montreal Cognitive Assessment (MoCA)(score of 16-23)
* Care partners will be included if they provide >10 hours of care/week
* Live in Baltimore City/County

Exclusion Criteria:

* Live in long term care setting

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Change in Function as assessed by the Katz Index of Independence in Activities of Daily Living | Baseline, 16 weeks, 32 weeks
  6 questions, each 1 point for a total score of 6. A score closer to 6 indicates high patient independence.
Change in Function as assessed by Lawton & Brody's assessment of Instrumental Activities of Daily Living Scale | Baseline, 16 weeks, 32 weeks
  The assessment contains 8 questions with answers that are either a score of 0 or 1. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women and 0 through 5 for men to avoid potential gender bias.
Change in Pain as assessed by the Brief Pain Inventory (Short Form) | Baseline, 16 weeks, 32 weeks
  The Brief Pain Inventory - Short Form is a 9 item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. The patient is asked to rate their worst, least, average, and current pain intensity, list current treatments and their perceived effectiveness, and rate the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life on a 10 point scale. For the 10 point scale, 0 indicated no pain and 10 indicates the worst imaginable pain.
Change in Depression as assessed by the Patient Health Questionnaire Depression Scale (PHQ-8) | Baseline, 16 weeks, 32 weeks
  The PHQ-8 contains 8 questions, with a 0-3 scale. A score of 10 or greater is considered major depression, 20 or more is severe major depression.
Change in caregiving burden as assessed by the Perceived Change Index Scale | 16 weeks, 32 weeks
  The Perceived Change Index Scale contains13 questions related to change in caregiver self-improvement wellbeing. Each rated on a scale of 1-5, 1 indicating much worse, 5 indicating improved a lot. The higher the overall score, the greater the improvement.
Change in Perceived Change in Function Scale Score | 16 weeks, 32 weeks
  14 questions related to perceived improvement in function. Scale of -2 (gotten much worse) to 2 (improved a lot). The higher the overall score, the greater the improvement.
Satisfaction at midpoint of intervention assessed by qualitative questions | 8 weeks
  Older Adult and Care Partner Satisfaction at midpoint of intervention assessed by qualitative questions. Qualitative questions will help us understand how best to tailor the intervention for the randomized control pilot.
Satisfaction at endpoint of intervention as assessed by qualitative questions | 16 weeks
  Older Adult and Care Partner Satisfaction at endpoint of intervention assessed by qualitative questions. Qualitative questions will help us understand how best to tailor the intervention for the randomized control pilot.
Level of Cognitive Impairment for eligibility as assessed by the Montreal Cognitive Assessment (MoCA) Blind/Telephone | Baseline
  Scoring for the Blind/Telephone assessment is out of 22. Score of 12-17 indicates Mild Cognitive Impairment/Early Stage Dementia and is the eligibility requirement for participation in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Szanton, PhD, RN, Principal Investigator — Johns Hopkins School of Nursing
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szanton SL, Wolff JW, Leff B, Thorpe RJ, Tanner EK, Boyd C, Xue Q, Guralnik J, Bishai D, Gitlin LN. CAPABLE trial: a randomized controlled trial of nurse, occupational therapist and handyman to reduce disability among older adults: rationale and design. Contemp Clin Trials. 2014 May;38(1):102-12. doi: 10.1016/j.cct.2014.03.005. Epub 2014 Mar 28. PMID 24685996